CLINICAL TRIAL: NCT03810807
Title: Phase 1 Study of Combination Dacomitinib and Osimertinib for Patients With Metastatic EGFR Mutant Lung Cancers
Brief Title: Study of Dacomitinib and Osimertinib for Patients With Advanced EGFR Mutant Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-411
Record Dates: First submitted 2019-01-17; First posted 2019-01-22 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Non-small Cell Lung Cancer
Keywords: Dacomitinib; Osimertinib; EGFR Mutant Lung Cancers; 18-411
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — dacomitinib; osimertinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dacomitinib and Osimertinib (Experimental): Patients will begin on combination dacomitinib and osimertinib at the prescribed doses.
  A cycle will be 28 days in duration. The study will use a standard 3+3 dose escalation design. Per MD discretion, telemedicine visits may be utilized for cycles where imaging is not collected, and physical exam, vital sign and labs collection will only be required concurrent with imaging visits.
  Interventions: Drug: Dacomitinib; Drug: Osimertinib

INTERVENTIONS:
Drug: Dacomitinib — Dose level 1 Dacomitinib, Dose level 2 Dacomitinib, Dose level 3 Dacomitinib. Three patients will need to be enrolled at each dose level and assessed for DLT for 1 full cycle (28 days for cycle 1) before dose escalation decision is made.
Drug: Osimertinib — Dose level 1, 2 and 3 Osimertinib 40mg daily. Three patients will need to be enrolled at each dose level and assessed for DLT for 1 full cycle (28 days for cycle 1) before dose escalation decision is made.

SUMMARY:
The purpose of this study is to test the safety of dacomitinib and osimertinib, at increasing doses, to find out what effects, if any, this combination of drugs has on people with metastatic EGFR mutant lung cancer that has not been treated with an EGFR TKI.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Advanced biopsy-proven metastatic non-small cell lung cancer
* Somatic activating mutation in EGFR in a tumor biopsy
* No prior EGFR inhibitor treatment (gefitinib, afatinib, erlotinib, dacomitinib, osimertinib) however, prior treatment with other chemotherapies are allowed
* Archival tissue available from a pre-treatment tumor biopsy or willing to undergo a tumor biopsy prior to study initiation.
* Measurable (RECIST 1.1) indicator lesion not previously irradiated
* Karnofsky performance status (KPS) ≥ 70%
* Age >18 years old
* Ability to swallow oral medication
* Agree to use effective methods of contraception from the time of screening until 3 months after treatment discontinuation (for males and females of child-bearing potential)
* Adequate organ function

  * AST, ALT ≤ 3 x ULN
  * Total bilirubin ≤1.5x ULN
  * Creatinine ≤ 1.5x ULN OR calculated creatinine clearance ≥ 60ml/min
  * Absolute neutrophil count (ANC) ≥ 1000 cells/mm^3
  * Hemoglobin≥9.0 g/dL
  * Platelets ≥100,000/mm^3

Exclusion Criteria:

* Pregnant or lactating women
* Any radiotherapy within 1 week of starting treatment on protocol.
* Any major surgery within 1 weeks of starting treatment on protocol.
* Any evidence of active clinically significant interstitial lung disease
* A mean QTc >470ms (Fridericia"s correction), clinically important arrhythmia, conduction or morphology of resting ECG (eg complete LBBB, 1st -3rd degree heart block, any factors that increase the risk of QTc prolongation or risk of arrhythmia)
* Cardiovascular disease or cerebrovascular disease, CVA or MI < 6 months prior to study enrollment, unstable angina, NYHA >Grade II CHF, or serious cardiac arrhythmia uncontrolled by medication or with the potential to interfere with protocol treatment
* History of pneumonitis or interstitial lung disease (ILD), drug induced ILD, radiation pneumonitits that required steroid treatment, and any evidence of clinically active ILD
* Serious chronic GI conditions associated with diarrhea
* Symptomatic, unstable brain metastases requiring escalating doses of steroids
* Continue to have unresolved > CTCAE grade 1 toxicity from any previous treatment

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-01-17 (Actual); Primary Completion 2025-12-15 (Actual); Study Completion 2025-12-15 (Actual)

PRIMARY OUTCOMES:
maximum tolerated dose | 1 year
  The MTD will be defined as the highest dose at which not more than 1/6 of the patients experience dose limiting toxicity (DLT). DLT is defined as any of the toxicity events described below that occurs within cycle 1 of treatment with the combination of dacomitinib and osimertinib.
Best overall response rate | 1 year
  Tumor response will be assessed using RECIST 1.1.The NCI Common Terminology Criteria for Adverse Events Version 5 (NCI-CTCAE) will be used to grade toxicities during the trial. Dose-limiting toxicities (DLT"s) are defined as any of the following events occurring during the first cycle of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Helena Yu, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.
Supporting Information: SAP, ICF

REFERENCES:
- [Derived] Poels KE, Schoenfeld AJ, Makhnin A, Tobi Y, Wang Y, Frisco-Cabanos H, Chakrabarti S, Shi M, Napoli C, McDonald TO, Tan W, Hata A, Weinrich SL, Yu HA, Michor F. Identification of optimal dosing schedules of dacomitinib and osimertinib for a phase I/II trial in advanced EGFR-mutant non-small cell lung cancer. Nat Commun. 2021 Jun 17;12(1):3697. doi: 10.1038/s41467-021-23912-4. PMID 34140482
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm